CLINICAL TRIAL: NCT01276964
Title: Protocol for the Determination of Menstrual Losses Using a System for the Quantitative Determination of Menses (Quantitative Evaluation of Menses [QUEM] Method) and Its Application to Healthy Women With Apparently Normal Cycles
Brief Title: Protocol for the Determination of Menstrual Losses in Healthy Women With Apparently Normal Cycles
Acronym: MEVA-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of L'Aquila (Other)
Collaborators: Casa Sollievo della Sofferenza IRCCS (Other); University of Palermo (Other)
Responsible Party: Principal Investigator, Guglielmo Mariani, Prof, University of L'Aquila
Other Study IDs: MEVA-1/2007
Record Dates: First submitted 2011-01-11; First posted 2011-01-14 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Validate QUEM Method; Quantitative Determination of Menses
Keywords: menses; quantitative determination of menstrual losses; kinetic definition of menses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Soiled oads and tampons, vacuum sealed are retained till their evaluation, they will be appropiately discharged after their analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1. Women in the fertile age: Healthy women in the fertile age (between 20-45 years) with apparently normal periods

SUMMARY:
Multicenter, observational, cross-over study intended to apply an easy and simple system for the quantitative determination of menstrual losses in women with apparently normal menses.The system adopted for the determination of menstrual losses, called QUEM (QUantitative Evaluation of Menses), is based on the collection of tampons and pads in standard bags which are readily vacuum sealed with a simple device for the whole of woman's period. The evaluation will be performed for the whole of one period and the analysis will be performed in comparison to the classical reference method, the Alkaline - Hematin Method, which is still considered the golden standard.

DETAILED DESCRIPTION:
The following is a multicenter, observational, cross-over study intended to apply an easy and simple system for the quantitative determination of menstrual losses in women with apparently normal menses. The problem of heavy periods is associated to an high social and physical morbidity rate; till now there are not routine methods available for the quantitative determination of menstrual discharge, some objective methods have been applied exclusively for research purposes because they are very difficult to perform. If we consider the scientific data available and the frequent application of inadequate procedures for the treatment of this problem, it seems essential to apply a practical system for the accurate quantitative determination of menses.

The system adopted for the determination of menstrual losses, called QUEM (QUantitative Evaluation of Menses), is based on the collection of tampons and pads in standard bags which are readily vacuum sealed with a simple device for the whole of woman's period. QUEM has already been validated in preliminary in vitro and ex vivo studies (both in healthy women and in women with CBDs), by comparing it with the gold standard, the Alkaline Haematin Method. A correlation coefficient close to 1 was obtained.

In the current study QUEM will be applied to at least 100 women in the fertile age (between 20 and 45 years) with apparently normal menses and a negative bleeding history. The evaluation will be performed for the whole of one period and the analysis will be performed in comparison to the classical reference method, the Alkaline - Hematin Method, which is still considered the golden standard. At the enrollment each woman will be tested for complete blood cells count and ferritin levels in order to exclude unknown menorrhagia. The bleeding history (bleeding score) will be performed by applying an international reference method, already validated for von Willebrand Disease type 1 (vWD1). The aim of the study is to make a "normal range" and validate the effective practicality of QUEM as a preliminary step to the clinical studies in patients suffering from menorrhagia and affected by hemorrhagic disorders.

The current study will involve many Italian and International Centers. All the needed materials and equipments will be provided by the Coordinator Centre; patients will be carefully informed about the objectives of the study and they will follow a short course illustrating the use and the characteristics of the method proposed (QUEM).

ELIGIBILITY:
Inclusion Criteria:

* Women in the fertile age (between 20-45 years), not assuming oral contraceptives from at least three months
* Referred normal menses .Use of the same brand of sanitary protection wear for the whole of the period.
* BMI between 18 and 30

Exclusion Criteria:

* Abnormal Bleeding Score
* Positive gynecological history of fibroids, polyps or malignancy
* Treatment with anti-coagulants, antifibrinolytics, non steroidal anti-inflammatory agents
* Use of oral contraceptives in past three months
* Use of intrauterine devices (IUDs) in past three months .Hgb levels <12 g/dl and Ferritin <25 ng/ml.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women in the fertile age with apparently normal cycles
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2007-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: mariasanta napolitano, md, Principal Investigator — univeristy of perugia, hospital of l'aquila; guglielmo mariani, md, Study Director — University of L'Aquila
Locations (3):
- Italy (3):
  - University of Palermo, Palermo, Italy
  - Casa Sollievo Della Sofferenza Irccs, San Giovanni Rotondo, Italy
  - University of L'Aquila, L’Aquila

REFERENCES:
- See also: The official site of Italian Society of Obstetrics and Gynecology — http://www.sigo.it
- See also: Official site of the American Society of Obstetrics and Gynecology for women's healthcare physicians — http://www.acog.org